CLINICAL TRIAL: NCT06298149
Title: Reach Through Equitable Implementation of Turtle Island Tales in American Indian Communities: Program Effectiveness
Brief Title: Reach Through Equitable Implementation of Turtle Island Tales
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Montana State University (Other)
Collaborators: National Institutes of Health (NIH) (NIH); University of Utah (Other); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2023-650-EXEMPT; 1U54CA280812-01 (NIH)
Record Dates: First submitted 2023-12-13; First posted 2024-03-07 (Actual); Last update posted 2025-10-15 (Actual); Status verified 2025-10

CONDITIONS: Obesity, Childhood; Obesity; Cancer
MeSH Terms: conditions — Pediatric Obesity; Obesity; Neoplasms

STUDY DESIGN:
Intervention Model Description: Each participating family will receive a monthly lesson targeting a healthy behavior (increase fruit/vegetable intake, decrease added sugar intake, increase physical activity, decrease sedentary/screen time, promote healthy sleep, and promote emotional regulation) over the course of one year.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Turtle Island Tales (Experimental): All participating families will receive a monthly lesson targeting a healthy behavior (increase fruit/vegetable intake, decrease added sugar intake, increase physical activity, decrease sedentary/screen time, promote healthy sleep, and promote emotional regulation) over the course of one year.
  Interventions: Behavioral: Turtle Island Tales

INTERVENTIONS:
Behavioral: Turtle Island Tales — All participating families will receive a monthly lesson targeting a healthy behavior (increase fruit/vegetable intake, decrease added sugar intake, increase physical activity, decrease sedentary/screen time, promote healthy sleep, and promote emotional regulation) over the course of one year.

SUMMARY:
Reach Through Equitable Implementation of Turtle Island Tales is a family-level obesity prevention intervention that aims to reinforce AI cultural values of family interaction and holistic wellness. The long-term objective of this research program is to increase the reach of existing evidence-based interventions (EBIs) for cancer and obesity prevention among American Indian (AI) families who live in persistent poverty census tracts.

DETAILED DESCRIPTION:
Turtle Island Tales is an obesity prevention program for AI families with young children (3-8 years) that was developed to address the gap in home-based, family wellness programs for this population. Substantial research as been conducted on the effectiveness of this program for participating families. The primary aim of the current project is to investigate community-engaged dissemination to improve the reach of Turtle Island Tales. Dissemination strategies will be undertaken in partnership with community leaders and/or local Supplemental Nutrition Assistance Program Education (SNAP-Ed) agents who will disseminate the program through existing Extension/SNAP-Ed delivery mechanisms (SNAP-Ed is commonly administered through Extension programs of land-grant universities). Turtle Island Tales was accepted as a SNAP-Ed eligible program in 2022. As such, the program will be administered as part of usual/typical SNAP-Ed delivery in participating communities and largely constitutes program evaluation.

The primary research question is: What is the reach of the evidence-based Turtle Island Tales wellness program intervention within AI communities? A secondary aim for this project is determining the effectiveness of Turtle Island Tales among participating families using program evaluation survey data obtained via SNAP-Ed program evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Residence in one of identified persistent poverty census tracts
* Person >18 years of age caring for a child 3-8 years old

Exclusion Criteria:

* Residence outside of identified persistent poverty census tracts
* Caregiver <18 years of age
* No child 3-8 years old living in household

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2028-04-30 (Estimated); Study Completion 2028-04-30 (Estimated)

PRIMARY OUTCOMES:
20-item Family Nutrition and Physical Activity Survey | one year
  Pre- and post-evaluation of effectiveness in behavioral outcomes including family-level questions targeting diet, physical activity, screen time, and sleep. The total score is used as the summary score, with a higher score indicating a more positive family home environment relative to health behaviors.

SECONDARY OUTCOMES:
Food insecurity screener | one year
  United States Department of Agriculture Household Food Insecurity 2-item screener: 1) "We worried whether our food would run out before we got money to buy more" and 2) "The food we bought just didn't last and we didn't have money to get more." An affirmative response ("Often True" or "Sometimes True") on either item is considered positive for food insecurity.
Mental Health screening | one year
  Two items from the validated Short Form-12 survey: 1) In the last month, how often have you felt that you were unable to control the important things in your life? and 2) In the last month, how often have you felt confident about your ability to handle your personal problems? Scores are summed, with a higher score being associated with more positive mental health status.

CONTACTS AND LOCATIONS:
Overall Officials: Emily Tomayko, PhD, Principal Investigator — Montana State University
Locations (1):
- Montana State University, Bozeman, Montana, United States

REFERENCES:
- [Background] Tomayko EJ, Prince RJ, Cronin KA, Parker T, Kim K, Grant VM, Sheche JN, Adams AK. Healthy Children, Strong Families 2: A randomized controlled trial of a healthy lifestyle intervention for American Indian families designed using community-based approaches. Clin Trials. 2017 Apr;14(2):152-161. doi: 10.1177/1740774516685699. Epub 2017 Jan 9. PMID 28064525
- [Background] Tomayko EJ, Webber EJ, Cronin KA, Prince RJ, Adams AK. Use of Text Messaging and Facebook Groups to Support the Healthy Children, Strong Families 2 Healthy Lifestyle Intervention for American Indian Families. Curr Dev Nutr. 2021 May 17;5(Suppl 4):32-39. doi: 10.1093/cdn/nzaa110. eCollection 2021 Jun. PMID 34222765
- [Background] Berns RM, Tomayko EJ, Cronin KA, Prince RJ, Parker T, Adams AK. Development of a Culturally Informed Child Safety Curriculum for American Indian Families. J Prim Prev. 2017 Apr;38(1-2):195-205. doi: 10.1007/s10935-016-0459-y. PMID 27913907
- [Result] Tomayko EJ, Prince RJ, Cronin KA, Adams AK. The Healthy Children, Strong Families intervention promotes improvements in nutrition, activity and body weight in American Indian families with young children. Public Health Nutr. 2016 Oct;19(15):2850-9. doi: 10.1017/S1368980016001014. Epub 2016 May 23. PMID 27211525
- [Result] Tomayko EJ, Prince RJ, Cronin KA, Kim K, Parker T, Adams AK. The Healthy Children, Strong Families 2 (HCSF2) Randomized Controlled Trial Improved Healthy Behaviors in American Indian Families with Young Children. Curr Dev Nutr. 2018 Nov 16;3(Suppl 2):53-62. doi: 10.1093/cdn/nzy087. eCollection 2019 Aug. PMID 31453428
- See also: Turtle Island Tales — http://turtleislandtales.org/aboutus